CLINICAL TRIAL: NCT04420026
Title: Study of the Contribution of Automatic Image Fusion of a Cone-beam CT Volume With Ultrasound During Percutaneous Ablation Treatment of Hepatic Tumors
Brief Title: Study of Automatic Image Fusion of a CT Volume With Ultrasound During Percutaneous Ablation Treatment of Hepatic Tumors
Acronym: IAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190581; 2019-A02524-53 (Registry Identifier: Registry ID: IDRCB)
Record Dates: First submitted 2020-05-04; First posted 2020-06-09 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: ablation; cone-beam CT volume; ultrasonography
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Hepatocellular tumours
  Interventions: Radiation: Interact Active Tracker

INTERVENTIONS:
Radiation: Interact Active Tracker — Interact Active Tracker, allowing the automation of the fusion between a CBCT and ultrasound imaging

SUMMARY:
The automatic fusion of the ultrasound with a cone-beam CT volume will guide the positioning of the electrodes, despite the visibility of the tumor in ultrasound, in patients treated with irreversible electroporation in the interventional radiology room at Avicenna Hospital for hepatocellular carcinoma (HCC). The objective is to evaluate the primary success rate of the automatic cone-beam CT fusion procedure and ultrasound, regardless of the tumor's visibility status in ultrasound.

DETAILED DESCRIPTION:
Percutaneous removal of hepatic tumours allows curative treatment using a range of techniques such as radiofrequency ablation, microwave, cryoablation or, more recently, irreversible electroporation. These treatments require the introduction of one or more electrodes into or around the areas to be treated. This insertion phase requires that the practitioner has a means of continuously visualizing the area to be treated and the position of the electrodes.

The reference modality for the treatment of hepatic tumours by ablation is ultrasound. The scanner is the conventional alternative recommended in case of invisibility of the target in ultrasound.

When the target is not clearly visible in ultrasound, advanced multimodal image fusion applications can allow the practitioner to overcome this difficulty. This fusion is made possible by tracking the movement of the ultrasound probe in relation to the patient using an electromagnetic navigation system, and by alignment between the ultrasound system and the fused volume.

This alignment can be done manually or automatically using a specific marker placed on the patient's skin, called an "Active Tracker".

The "INTERACT Active Tracker" functionality will also simplify the registration process by providing automatic pre-registration.

The purpose of this study is to prospectively evaluate the primary success of patients treated at Avicenna Hospital for HCC by irreversible electroporation using this fusion technique. The hypothesis of the study is that this image fusion makes it possible to improve the location of the lesions to be treated and to allow treatment by percutaneous ablation of lesions that are not very visible under ultrasound alone.

This study will also assess the time and accuracy savings when an automatic fusion solution between ultrasound and cone-beam (CB) CT is used, compared to manual alignment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient treated at Avicenna Hospital for HCC by irreversible electroporation (IRE)
* Patient whose tumor treatment requires the use of fusion tools with CBCT imaging at the beginning of the procedure
* Patients with a scheduled follow-up examination 1 month after the ablation procedure by irreversible electroporation (IRE)
* Patient who has understood the information and agreed to participate in this research by signing the consent form
* Patient affiliated to a social security system or entitled person

Exclusion Criteria:

* Patients with a history of allergy to iodinated contrast material
* Patients with MRI contraindications
* Patients with a history of allergy to contrast material containing gadolinium
* Pregnant or breastfeeding women
* Patients under the protection of justice
* Patients unable to understand research information in an informed manner
* Participation in another interventional therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of the primary success rate of percutaneous ablation treatment with IRE of hepatic tumors, as a function of the ultrasound visibility of the tumor, when using automatic CT cone-beam fusion and ultrasound | At 1 month on post-operative imaging
  Primary success is assessed on the control MRI or CT performed one month after the first IRE (Irreversible Electroporation) ablation procedure targeting a given tumor. It is defined by the absence of visible recurrence at 1 month on post-operative imaging. In the case of a partial response, a % of active tumor will be evaluated.

SECONDARY OUTCOMES:
Evaluate the time savings when using "INTERACT Active Tracker" allowing automatic alignment of the CBCT volume with ultrasound | The day of the operation
  The ultrasound visibility of the tumor is evaluated by an ordered discrete variable defined as follows:
  0: Not identifiable with or without merging
  1. identifiable with the help of fusion, tumor boundaries are poorly defined
  2. identifiable with the help of fusion, the limits of the tumour are clearly visible
  3. identifiable without fusion, tumor boundaries are poorly defined
  4. identifiable without fusion, the limits of the tumour are clearly visible
Evaluate the time saved by using "INTERACT Active Tracker" allowing automatic alignment of the CBCT volume with ultrasound compared to the manual alignment procedure performed on a series of patients treated when the new function was not available. | The day of the operation
  Time is measured from the moment the entire volume is loaded onto the ultrasound scanner. The stopwatch is stopped when the operator declares himself satisfied with the adjustment
Evaluate the confidence gain associated with the use of ultrasound fusion. | The day of the operation
  The confidence gain associated with the use of ultrasound fusion is assessed by noting the number of non-visible or non-localizable tumors in ultrasound alone that can be identified through fusion.
Evaluate the accuracy of the automatic alignment judged on the ultrasound measurement of the distance from the center of the target seen in ultrasound to that segmented on the pre-therapeutic pour Cone Beam Computed Tomography (CBCT). | The day of the operation
  The accuracy of the automatic alignment judged on the ultrasound measurement of the distance from the center of the target seen in ultrasound to that segmented on the pre-therapeutic CBCT is evaluated by comparison with the accuracy of the manual alignment recorded on a series of patients treated when the new function was not available
Evaluate the percentage of procedures for which similarity points must be added due to an initial delay in automatic merging that the operator considers too long. | The day of the operation
  The percentage of procedures for which similarity points must be added due to an initial delay of the automatic merge considered too long by the operator is evaluated in comparison with the historical series (manual alignment, when the new function was not available).
Evaluate the failure rate of the Interact Active Tracker automatic alignment. | The day of the operation
  If the operator is not satisfied with the automatic registration between the CBCT and ultrasound, the number of similarity point(s) to be placed and the time required to make this adjustment will be recorded
Evaluate the secondary and third-party therapeutic effectiveness rate of the procedures. | The day of the operation
  The failure rate of the Interact Active Tracker automatic alignment is evaluated by the number of procedures where this function is not functional for any reason. Throughout the procedure, the number of times the operator will have to correct the alignment with new anatomical landmarks will be counted. Any failure of the automatic merge will be recorded.
For incomplete responses, estimate the percentage of active tumour (enhanced by contrast material). | One month after the ablation
  The secondary and third-party therapeutic effectiveness rate of the procedures is defined by the number of cases in which two or three ablation procedures will be required to achieve a complete MRI response within one month of the last ablation session. For each tumour, the number of ablation procedures required to achieve a complete MRI response within one month of the last ablation session will be recorded. For patients requiring more than one treatment, only treatments performed over the duration of the study should be included.
Assess the complication rate. | The day of the ablation
  The complication rate is evaluated by the Dindo-Clavian classification so complication will be recorded and classified
Evaluate the global survival at 12 months | 12 months after the ablation
  Overall survival at 12 months. It will be collected by consulting medical records based on the recorded dates of the last visits, images...

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Mr SEROR, PhD, Principal Investigator — Assistance Publique - Hôpitaux Paris
Locations (1):
- SERROR, Bobigny, France

REFERENCES:
- [Background] Nault JC, Sutter O, Nahon P, Ganne-Carrie N, Seror O. Percutaneous treatment of hepatocellular carcinoma: State of the art and innovations. J Hepatol. 2018 Apr;68(4):783-797. doi: 10.1016/j.jhep.2017.10.004. Epub 2017 Oct 13. PMID 29031662
- [Background] Yu H, Burke CT. Comparison of percutaneous ablation technologies in the treatment of malignant liver tumors. Semin Intervent Radiol. 2014 Jun;31(2):129-37. doi: 10.1055/s-0034-1373788. PMID 25071303
- [Background] Monfardini L, Orsi F, Caserta R, Sallemi C, Della Vigna P, Bonomo G, Varano G, Solbiati L, Mauri G. Ultrasound and cone beam CT fusion for liver ablation: technical note. Int J Hyperthermia. 2018;35(1):500-504. doi: 10.1080/02656736.2018.1509237. Epub 2018 Sep 11. PMID 30204007
- [Background] Lee LH, Hwang JI, Cheng YC, Wu CY, Lee SW, Yang SS, Yeh HZ, Chang CS, Lee TY. Comparable Outcomes of Ultrasound versus Computed Tomography in the Guidance of Radiofrequency Ablation for Hepatocellular Carcinoma. PLoS One. 2017 Jan 9;12(1):e0169655. doi: 10.1371/journal.pone.0169655. eCollection 2017. PMID 28068369
- [Background] Cornelis FH, Korenbaum C, Ben Ammar M, Tavolaro S, Nouri-Neuville M, Lotz JP. Multimodal image-guided electrochemotherapy of unresectable liver metastasis from renal cell cancer. Diagn Interv Imaging. 2019 May;100(5):309-311. doi: 10.1016/j.diii.2019.01.001. Epub 2019 Jan 26. No abstract available. PMID 30691970
- See also: Minimally Invasive Treatments for Liver Cancer, Updates in Liver Cancer. Nicolas Cardenas, Rahul Sheth and Joshua Kuban. — https://www.intechopen.com/books/updates-in-liver-cancer/minimally-invasive-treatments-for-liver-cancer